CLINICAL TRIAL: NCT07274124
Title: Comparison of the Effects of Pain Neuroscience Education and Vagus Nerve Stimulation on Recovery in Individuals With Rheumatoid Arthritis
Brief Title: Pain Neuroscience Education and Vagus Nerve Stimulation on Recovery in Individuals With Rheumatoid Arthritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Simay Akdemir, MSc. Phd Candidate, Lecturer Physical Therapist, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-7253
Record Dates: First submitted 2025-11-19; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Rheumatic Diseases; Rheumatoid Arthritis (RA)
Keywords: rheumatoid arthritis; pain neuroscience education; vagal nerve stimulation; exercise
MeSH Terms: conditions — Rheumatic Diseases; Arthritis, Rheumatoid; Motor Activity | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: The study will be conducted using a randomized, controlled, prospective design. Thirty-six individuals diagnosed with RA at the Department of Rheumatology at Cerrahpaşa Faculty of Medicine Hospital will be included in the study. Following the physician referral, individuals who meet the inclusion criteria will be divided into three equal groups (12 in each), by using block randomization by the "randomizer.org" website, and the number of cases will be calculated using the "GPower" application. Demographic information will be collected before the study begins, and all participants will be informed in advance of the study's purpose, duration, and content, as well as the voluntary nature of their participation with an informed consent form. After the initial assessment, the intervention will last for 8 weeks and consist of three groups: "Pain Neuroscience Education-PNE + Structured Exercise," "Transauricular Vagus Nerve Stimulation-tVNS + Structured Exercise," and "Structured Exercise."
Who Masked: Participant
Masking Description: Patients who are taken into one of the three intervention groups will not have any idea or information about the interventions being performed in other groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pain Neuroscience Education + Structured Exercise (Experimental): The PNE method will be applied simultaneously with exercise. Training will begin after the first session, which includes a face-to-face assessment. On the first day, a PowerPoint presentation will introduce the patient about pain anatomy, physiology, factors affecting pain, and central and peripheral sensitization. The topic of pain will be introduced, and the patient will be informed about the process. Pain mechanisms will be reviewed using video explanations, visual aids, and animations, information will be provided on what physical activity is and its effects on pain, patients will be asked their opinions on exercise, suggestions for physical daily, living activities will be given such as increasing activity, using stairs, limiting screen time type of suggestions will be thought to the patient and the patient's wishes and goals will be questioned in the further sessions. Each session will last 30 minutes and 16 education sessions will be completed in total.
  Interventions: Other: Pain Neuroscience Education; Other: Structured Exercises
- Vagal Nerve Stimulation + Structured Exercise (Experimental): Will be applied with the non-invasive taVNS-Research (tVNS®) device, which is the only safe auricular vagus stimulation device approved by the Ministry of Health in Türkiye and is used in various diseases such as headache, epilepsy, and fibromyalgia. Electrodes will be placed on the left auricular cavum conchae using two carbon-impregnated silicone electrodes to reduce the risk of cardiac side effects. Vagal nerve stimulation will be administered twice a week for 8 weeks, with a total of 16 supervised sessions. During this period, the home exercise intervention that patients are asked to perform will continue. Following the initial evaluation, the exercises will be taught to the patient, and the first nerve stimulation session will be performed. Current intensity will be adjusted according to the patient tolerance-threshold value, and this value will be recorded for each session.
  Interventions: Other: Vagal Nerve Stimulation; Other: Structured Exercises
- Structured Exercise (Active Comparator): The Structured exercise intervention, specifically for individuals with RA and designed to target painful areas, will be implemented in the form of home exercises for all three groups, twice a week for 8 weeks. The exercise program will primarily consist of warm-up, basic exercise, and a cool-down period. Aerobic, strengthening, flexibility, breathing, and hand exercises will be planned based on EULAR recommendations. The warm-up period will begin with flexibility and range of motion exercises, followed by calisthenic and therapeutic endurance and strengthening exercises, and the session will ended with diaphragmatic breathing and hand exercises during the cool-down period. Additionally, walking activity will be recommended for at least two days per week.
  Interventions: Other: Structured Exercises

INTERVENTIONS:
Other: Pain Neuroscience Education — Many sources in the literature draw attention to patient education as the first stage of treatment and the most common educational technique that focuses on the perception, mechanism and modulation of pain is known as Pain Neuroscience Education (PNE). Patients in this group will take educational sessions about the pain, facilitators of pain, the factors affecting the pain perception and how to deal with chronic pain in rheumatoid arthritis with the help of power point presentations, animation videos, pictures and drawings. Intervention will last for 8 weeks, 2 times per week, in total 16 sessions will be completed. Each session will last 30 minutes in average and at the same time, patients will be advised to perform the given home exercises for 2 times per week. Assessments will be performed before and after the intervention.
  Arms: Pain Neuroscience Education + Structured Exercise
Other: Vagal Nerve Stimulation — Vagus nerve (cranial nerve X) is the longest and most widely distributed cranial nerve containing sensory, motor, and parasympathetic fibers. It plays an important role in the regulation of cardiovascular, respiratory, immune, endocrine, and autonomic systems, as well as homeostasis. Participants with rheumatoid arthritis will be taken into stimulation sessions for 2 times per week for continuous 8 weeks. Assessments will be performed before study and after the 16 sessions are completed. Since the literature has missing knowledge about the effects of Vagal nerve stimulation in rheumatoid arthritis, the results will highlight the effects on pain and inflammatory markers in this population. Current will be given from the left ear/transauricular area to prevent the side effects in the sessions.
  Arms: Vagal Nerve Stimulation + Structured Exercise
Other: Structured Exercises — Structured exercise planned in this study is based on the principles and suggestions of EULAR, by consisting warm-up, basic exercise and warm up sessions by combining different exercise types like aerobic, strengthening flexibility, breathing and definitely by including hand specific exercises. Participants in all three groups will be educated in the first session about the exercises to prevent wrong application and injuries. Afterwards, all groups will continue to their exercises at the home setting. An exercise diary will be asked from patients to control if they continue to their exercises regularly for 2 times for 8 weeks.

SUMMARY:
In the context of this randomized controlled study, patients who are diagnosed with Rheumatoid arthritis in Cerrahpaşa Faculty of Medicine Hospital, will be taken into a rehabilitation program by a qualified physiotherapist to improve their pain, pain perception, inflammatory markers and quality of life, with one of the pain neuroscience education, vagal nerve stimulation and traditional exercise interventions. The results of each intervention method will be analyzed and compared at the end of the 8 weeks study protocol.

DETAILED DESCRIPTION:
Pain, a complex and multifaceted experience, is the most common symptom observed in inflammatory arthritis. In addition to pathological events such as inflammation and tissue infection, various personal, social, and behavioral factors such as illness beliefs, mood, behavior, avoidance, sleep disturbance, and daily rest and activity status also contribute to pain and pain perception. According to the 2018 EULAR recommendations, the principles of pain management methods are based on a patient-centered care and social assistance models of rehabilitation. According to PNE, the primary cause of chronic pain is not an organ or tissue damage, but rather over activation of the central nervous system and central sensitization and the goal is to reduce CNS activation, minimize fear of movement, and increase pain tolerance, thereby supporting exercise participation. Based on the biopsychosocial model, this method aims to reduce movement and illness avoidance behavior by reshaping pain perception. It is typically presented to patients through one-on-one or group meetings, phone calls, or visual brochures. Another effective method on the indicated pain related symptoms is known as Vagal nerve stimulation. Neural regulation can be achieved by vagal nerve stimulation, which is related to the pain-processing pathways of the brain, or pain reduction can be achieved indirectly through the anti-inflammatory effect it creates. While studies in the literature on VNS mostly focus on individuals with chronic pain, fibromyalgia, abdominal pain, and headache, there are few studies on rheumatoid arthritis. Besides no studies have examined the effects of PNE. This research points to a significant deficiency in pain perception, awareness, and control in individuals with RA. Based on this information, the aim of this study was to examine the effects of pain neuroscience training and vagal nerve stimulation on healing parameters in individuals with rheumatoid arthritis and to compare the results in terms of their superiority.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who were diagnosed with RA at least one year ago,
* Ages of 18 and 65,
* Have been experiencing pain for three months or more,
* Score 24 or higher on the Mini Mental State Examination (MMSE), and can follow instructions will be included in the study.

Exclusion Criteria:

* Individuals under 18 years of age,
* Reporting acute pain or pain from injury,
* Having a history of surgery within the last year,
* Having a score of <24 on the MMSE,
* Having any of the cerebrovascular disease, cardiovascular disease, symptomatic coronary artery disease, myocardial infarction, congestive heart failure, or uncontrolled hyper/hypotension,
* History of vagotomy surgery, or having an implanted electrical/neurostimulator device will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Pain Catastrophizing Scale | 8 weeks
  13-item questionnaire, based on personal feedback, assesses the severity of patients' reactions to pain on a scale of 0-4. The validity and reliability of the questionnaire in Turkish has been established.
Disease Activity Score-28 (DAS28) | 8 weeks
  Assesses disease activity in 28 different joints. Blood draws will be performed by a specialist physician who diagnoses patients, conducts regular checkups, and then refers suitable patients to a physical therapist. A score below 2.6 indicates the disease is in remission; scores between 2.6 and 3.1 indicate low disease activity; scores between 3.1 and 5.1 indicate moderate disease activity; and scores above 5.1 indicate high disease activity.

SECONDARY OUTCOMES:
Demographic Information Form | At the beginning only
  The patient's personal information, medical treatment history, current lifestyle, and exercise habits will be inquired about using a form specifically designed for the specific disease.
Mcgill Pain Questionnaire Short Form | 8 weeks
  Developed by Melzack in 1987, the questionnaire assesses chronic pain in three sections: pain characteristics, severity, and intensity, has also been validated in Turkish and is recommended for use in rheumatological patients. The Turkish validation of the questionnaire was conducted by Yavuz et al. in 2007, and it was found to be valid in Turkish. Higher score indicates severe pain severity.
Pain Algometry | 8 weeks
  The pressure pain threshold (PPT), defined as the minimum pressure stimulus applied to elicit pain, is suitable for measuring pain in RA. Pain thresholds will be measured using an algometer at the third metacarpophalangeal (MCP) joints, the wrist, and the most inflamed joints.
Pain Coping Inventory | 8 weeks
  Indicates how frequently patients use behavioral and cognitive methods to cope with pain. The questionnaire, consisting of 6 subscales (active and passive), inquires about patients' orientations during painful situations. Items are scored on a 4-point Likert scale, with 1 being the least frequent use of pain management measures and 4 being the most frequent.
Tampa Kinesiophobia Scale | 8 weeks
  Published in 1995 to measure fear of movement and re-injury, the questionnaire consists of 17 items. Questions address areas such as fear of re-injury and avoidance of movement. A score of 17 is the lowest possible score, and indicates no kinesiophobia or negligible.
Bristol Rheumatoid Arthritis Multidimensional Fatigue Questionnaire | 8 weeks
  Examines the various dimensions of the effects of RA on fatigue. It was developed in 2010. The questionnaire consists of four subcategories: physical fatigue in the last 7 days, fatigue in activities of daily living, and cognitive and emotional fatigue. Patients receive scores between 0 and 70 on the 20-question questionnaire, with higher scores indicating higher fatigue.
Pittsburgh Sleep Quality Scale | 8 weeks
  19-item scale questions subjective sleep quality over the past month. The total score ranges from 0 to 21, with a higher score indicating poor sleep quality. A Turkish version of the scale is available and is used in rheumatological diseases.
Rheumatoid Arthritis Quality of Life Scale | 8 weeks
  30-item scale, with valid and reliable Turkish versions, is a published quality of life questionnaire specific to rheumatoid arthritis. Higher scores indicate lower quality of life.
Upper and Lower Extremity Goniometry and Circumference Measurements | 8 weeks
  To examine the relationship between pain and joint range of motion, goniometry measurements will be taken at the four most commonly affected areas: the atlantoaxial joint, shoulder joint, wrist joint, and ankle with the degree of movement.
  Circumference measurements will be taken at the hand, finger, and ankle to assess inflammation in the centimeter measures.
Multiple Choice Questions and Answers | 8 weeks
  Participants in the PNE group will be asked to answer 10 multiple-choice questions covering the presentation topics. This will provide information about the level of understanding of the information presented within the PNE group and its impact on the pain questionnaires, according to the score they take out of the total score of 100.

CONTACTS AND LOCATIONS:
Overall Officials: Simay AKDEMİR, MSc. Phd Candidate/Lec., Principal Investigator — İstanbul University-Cerrahpaşa
Locations (1):
- Cerrahpaşa Faculty of Medicine Hospital, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No